CLINICAL TRIAL: NCT02064517
Title: Randomized Comparative Test Multicentric, Forward-looking Single-blind, Between a Reference Technique and an Innovative Technic.
Brief Title: Treatments of the Necrosed Immature Teeth (REV)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lake of inclusion
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29BRC12.0131; Revascularisation pulpaire
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Clinical and Radiographic Success in 24 Months
Keywords: Necrosed Immature monoradicular Teeth , Revascularisation pulpar, MTA apical barrier, Clinical and radiographic success

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional technique (Placebo Comparator): Apical MTA barrier
  Interventions: Device: MTA
- Revascularisation pulpaire (Experimental): hydroxide of calcium
  Interventions: Device: Hydroxide of calcium

INTERVENTIONS:
Device: MTA — Creation of a barrier apicale in the MTA
  Arms: Conventional technique
Device: Hydroxide of calcium — Revascularisation pulpaire with some hydroxide of calcium
  Arms: Revascularisation pulpaire

SUMMARY:
Estimate if the technique of revascularisation pulpaire (with some hydroxide of calcium) allows to obtain a better forecast of preservation of the tooth without complication than the conventional technique with the creation of an apicale barrier in the MTA in 24 months.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting one or monoradicular immature definitive several teeth ( open apex) with a pulpar necrosis,
* 6-year-old patients in 17 years the parents(relatives) of which agree to give a lit(enlightened) written consent or patients of more than 18 years old.

Exclusion Criteria:

* general order: any pathology or treatment(processing) dissuading a treatment(processing) endodontic (patients at risk of infectious endocarditis) or pulling(entailing) an immunosuppression (diabetes, HIV, immunosuppresseurs treatments(processings) post-transplant, long-term corticoids, chemotherapies), allergy known about the used, antecedent products of cervico-facial radiotherapy, presenting subject of the communications problems, the pregnancy and the feeding.
* local order: generalized periodontal disease or superior located(localized) periodontal pocket in 3mm, crack or fracture(split) radiculaire, radiculaire reduction of the necrosed immature tooth

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Followed in 24 months | 24 months
  Clinical and radiological follow-up in 24 months

SECONDARY OUTCOMES:
Clinical and radiographic success | 3-6 months
  Clinical and radiographic success in 3 months, 6 months, 12 months and 18 months
Return of the pulpaire sensibility | 3-6 months
  Test of thermal and electric sensibility
Obtaining of a closure apicale and of an increase of length and thickness of radiculaires walls | 3-6 months
  radiographies with an angulateur and an abutment of repositioning
Appearance of complications (dyschromie dental) | 3-6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest - Pôle Organe des Sens, Brest
  - Hôtel Dieu, Nantes
  - CHU de Rennes, Rennes